CLINICAL TRIAL: NCT05693571
Title: Engagement and Depression in Adolescents and Young Adults With CHildhood-Onset Systemic Lupus
Brief Title: Engagement in CHildhood-Onset Systemic Lupus
Acronym: ECHOS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Childhood Arthritis and Rheumatology Research Alliance (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-14314; K23AR080803 (NIH)
Record Dates: First submitted 2022-12-05; First posted 2023-01-23 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Lupus Erythematosus, Systemic; Depression
Keywords: Engagement in care; Mobile health
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Valera Pilot Study (Experimental): All participants in the open-label pilot study will be provided with the Valera smart phone application and online care manager dashboard
  Interventions: Behavioral: Valera Smart Phone Application and Care Manager Dashboard

INTERVENTIONS:
Behavioral: Valera Smart Phone Application and Care Manager Dashboard — Valera mobile health application will provide educational materials around mental health and Systemic Lupus Erythematosus (SLE) and the ability to connect to a SLE care team via a care manager.

SUMMARY:
The goal of this observational (Aim 1) and pilot study (Aim 2) is to better understand how depression symptoms may contribute to how well adolescent and young adults with lupus follow-up with their lupus clinical care. The main questions the overall study attempts to answer are:

1. Whether anhedonia (a core symptom of depression) predicts disengagement in care
2. Whether a patient-tailored mobile health application built to improve both engagement in care and depression symptoms will be feasible and acceptable to adolescents and young adults with lupus.

Participants with systemic lupus, ages 15-24 from the Bronx, New York will be asked to complete questionnaires; some will be asked to participate in focus groups to help adapt the mobile health app; participants will also be invited to join a pilot study to try the mobile health app for 6 months and answer questionnaires to document the experience.

DETAILED DESCRIPTION:
This registration is exclusive to the pilot study (Protocol Aim 2). The primary objective of Aim 2 is to assess the feasibility and acceptability of an adapted Valera application (app) in adolescents and young adults (AYA) with childhood-onset systemic lupus erythematosus (cSLE). As a part of Aim 1 (not a component of this registration), using a recognized patient-engaged methodology, "ADAPT-ITT"22, the study team will iteratively adapt and test the content and utilities of the app for cSLE AYA. During the 6-month pilot study which constitutes Aim 2, the investigator team will examine feasibility and acceptability through mixed-methods. Feasibility and acceptability will be assessed via app use and validated feasibility and acceptability of intervention measures.

ELIGIBILITY:
Inclusion Criteria:

* Participants 15-25 years old meeting American College of Rheumatology (ACR) Revised SLE Classification Criteria and/or European League Against Rheumatism/ACR Classification Criteria and/or 2012 SLE International Collaborating Clinic Criteria and followed at the Children's Hospital at Montefiore.
* Must be diagnosed with SLE before 19 years of age (based on Childhood-onset systemic lupus erythematosus (cSLE) definition)

Exclusion Criteria:

* Non-Spanish or non-English speaking
* Participants anticipating transitioning to an outside rheumatologist for lupus care within the period of study follow-up
* Current psychotic disorders. However, attention-deficit/hyperactivity disorder, anxiety disorders, obsessive-compulsive disorder, posttraumatic stress disorder, eating disorders, and substance abuse disorders are not uncommon among adolescents and young adults (AYA) and will be allowed. Suicidal ideations (SI) and self-injurious acts (cutting) are common in depression and will be allowed (defined as passive SI).

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Application Utilization | 6 months
  Feasibility of the Valera health application will determined by the percentage of participants who utilize the Valera platform. Participants with repeated (i.e., ≥ 2) log-ins to both the care management and educational platforms will be considered users. A successful target percentage of ≥ 80% of enrolled participants logging into the care plan on the application and utilizing the messenger system at least twice during the 6-month pilot will be considered highly feasible.
Feasibility of the Intervention Measure (Participant Rating of Application Feasibility) | 6 months
  Feasibility of the Intervention Measure (FIM) will be assessed by participant rating of application feasibility via administration of a 4-item questionnaire at the end of the pilot study. Responses to each of the 4 questions will be evaluated on a 5-point scale as follows: (1 = "Completely disagree", 2 = "Disagree", 3 = "Neither agree nor disagree", 4 = "Agree", 5 = "Completely agree"). A higher aggregate score denotes a more favorable participant rating of feasibility of the application.

SECONDARY OUTCOMES:
Acceptability of the Intervention Measure (Participant Rating of Application Acceptability) | 6 months
  Acceptability of the Intervention Measure (AIM) will be assessed by participant rating of application acceptability via administration of a 4-item questionnaire at the end of the pilot study. Responses to each of the 4 questions will be evaluated on a 5-point scale Response (1 = "Completely disagree", 2 = "Disagree", 3 = "Neither agree nor disagree", 4 = "Agree", 5 = "Completely agree"). A higher aggregate score denotes a more favorable participant rating of the application. For purposes of this study a group mean score of ≥4 (representing "Agree" or "Completely agree") across the 4 items in ≥80% or participants will be an indicator of Acceptability.

OTHER OUTCOMES:
Engagement in Care - Number of participants with one or more lupus visits | 6 months
  Engagement in Care will be defined by the number of participants who have completed at least 1 clinical cSLE visit during the 6-month pilot window.
Change in SLE disease activity - patient reported | 3 months
  Change from baseline in patient reported lupus disease activity will be assessed using the SLE Activity Questionnaire (SLAQ). The SLAQ is an assessment tool which consists of 24 questions related to the severity and symptoms of lupus over the prior 30 days rated on a Likert-like scale ranging from 0 ("No problem") to 3 ("Severe") as well as a single Patient Global Assessment question about presence of lupus activity disease activity over the prior 30 days scored on a scale of 0 ("No activity") to 10 ("Most activity"). For purposes of this study change from baseline is being assessed such that a positive value signifies increased lupus disease activity from baseline and a negative value signifies decreased lupus disease activity from baseline.
Change in SLE disease activity - patient reported | 6 months
  Change from baseline in patient reported lupus disease activity will be assessed using the SLE Activity Questionnaire (SLAQ). The SLAQ is an assessment tool which consists of 24 questions related to the severity and symptoms of lupus over the prior 30 days rated on a Likert-like scale ranging from 0 ("No problem") to 3 ("Severe") as well as a single Patient Global Assessment question about presence of lupus activity disease activity over the prior 30 days scored on a scale of 0 ("No activity") to 10 ("Most activity"). For purposes of this study change from baseline is being assessed such that a positive value signifies increased lupus disease activity from baseline and a negative value signifies decreased lupus disease activity from baseline.
Change in SLE disease activity - clinically assessed | 3 months
  Change from baseline in clinically assessed lupus disease activity as defined by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI 2K). SLEDAI-2K is a scoring system based on the (binary) presence or absence of 24 descriptors in nine organ systems assessed over the preceding 30 days. Each of the descriptors has a weighted score and the total score of SLEDAI-2K is the sum of all 24 descriptor scores (range 0-105). For purposes of this study change from baseline is being assessed such that a positive value represents increased SLE disease activity relative to baseline based on the SLEDAI 2K and a negative value represents decreased SLE disease activity relative to baseline based on the SLEDAI 2K.
Change in SLE disease activity - clinically assessed | 6 months
  Change from baseline in clinically assessed lupus disease activity as defined by the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI 2K). SLEDAI-2K is a scoring system based on the (binary) presence or absence of 24 descriptors in nine organ systems assessed over the preceding 30 days. Each of the descriptors has a weighted score and the total score of SLEDAI-2K is the sum of all 24 descriptor scores (range 0-105). For purposes of this study change from baseline is being assessed such that a positive value represents increased SLE disease activity relative to baseline based on the SLEDAI 2K and a negative value represents decreased SLE disease activity relative to baseline based on the SLEDAI 2K.
Change in Depression symptom severity - Beck Depression Inventory-II (BDI-II) | 3 months
  Change from baseline in patient reported depression symptoms severity as defined by Beck Depression Inventory-II (BDI-II). This questionnaire consists of a 21-item self-reporting inventory answered by the participant based on a 4-point scale of increased severity of depression symptoms over the prior 2-week period. The BDI score is based on a 4-point scale, with 0 indicating no impairment and 3 indicating severe impairment for a possible overall scoring range of 0-63. For purposes of this study change from baseline is being assessed such that a positive value represents increased depression symptom severity relative to baseline based on BDI-II and a negative value represents decreased depression symptom severity relative to baseline based on the BDI-II.
Change in Depression symptom severity - Beck Depression Inventory-II (BDI-II) | 6 months
  Change from baseline in patient reported depression symptoms severity as defined by Beck Depression Inventory-II (BDI-II). This questionnaire consists of a 21-item self-reporting inventory answered by the participant based on a 4-point scale of increased severity of depression symptoms over the prior 2-week period. The BDI score is based on a 4-point scale, with 0 indicating no impairment and 3 indicating severe impairment for a possible overall scoring range of 0-63. For purposes of this study change from baseline is being assessed such that a positive value represents increased depression symptom severity relative to baseline based on BDI-II and a negative value represents decreased depression symptom severity relative to baseline based on the BDI-II.
Change in Depression symptom severity - Patient Health Questionnaire-9 (PHQ-9) | 3 months
  Change from baseline in patient reported depression symptoms severity will be assessed using the PHQ-9. The PHQ-9 is a 9-item self-reporting inventory answered by the participant related to the severity of their depression symptoms over the prior 2-week period. As a severity measure, responses to the PHQ-9 questions are scored on a 4-point scale ranging from 0 ("Not at all") to 3 ("Nearly every day") and a composite score is summed from the individual items. For purposes of this study change from baseline is being assessed such that a positive value represents increased depression symptom severity relative to baseline based on the PHQ-9 and a negative value represents decreased depression symptom severity relative to baseline based on the PHQ-9.
Change in Depression symptom severity - Patient Health Questionnaire-9 (PHQ-9) | 6 months
  Change from baseline in patient reported depression symptoms severity will be assessed using the PHQ-9. The PHQ-9 is a 9-item self-reporting inventory answered by the participant related to the severity of their depression symptoms over the prior 2-week period. As a severity measure, responses to the PHQ-9 questions are scored on a 4-point scale ranging from 0 ("Not at all") to 3 ("Nearly every day") and a composite score is summed from the individual items. For purposes of this study change from baseline is being assessed such that a positive value represents increased depression symptom severity relative to baseline based on the PHQ-9 and a negative value represents decreased depression symptom severity relative to baseline based on the PHQ-9.
Change in Perceived Stress | 3 months
  Change from baseline in patient reported perceived stress severity will be assessed using a Perceived Stress Scale 10 item questionnaire. Participants are asked to provide responses to each question based on their feelings and thoughts related to stressors over the prior month. Responses to the 10 items are scored on a 5-point scale ranging from 0 ("Never") to 4 ("Very Often") and a composite score is summed from the individual items. For purposes of this study change from baseline is being assessed such that a positive value signifies an increased level of perceived stress relative to baseline and a negative value signifies a decreased level of perceived stress from baseline.
Change in Perceived Stress | 6 months
  Change from baseline in patient reported perceived stress severity will be assessed using a Perceived Stress Scale 10 item questionnaire. Participants are asked to provide responses to each question based on their feelings and thoughts related to stressors over the prior month. Responses to the 10 items are scored on a 5-point scale ranging from 0 ("Never") to 4 ("Very Often") and a composite score is summed from the individual items. For purposes of this study change from baseline is being assessed such that a positive value signifies an increased level of perceived stress relative to baseline and a negative value signifies a decreased level of perceived stress from baseline.
Change in Self efficacy for medications and therapy | 6 months
  Change from baseline in self-efficacy will be assessed using the Patient Reported Outcome Measurement Information System (PROMIS) Self-efficacy treatment and medication questionnaire. This 26-item questionnaire measures patient confidence in taking medications and handling therapy in the context of potential challenges. Responses to each item are scored on a 5-point Likert-like scale ranging from 1 ("I am not at all confident") to 5 ("I am very confident"). Raw itemized scores are aggregated and transformed to a T-score using a linear transformation. The T-score is centered at 50 with a standard deviation of 10 such that 50 is considered average. Higher scores (e.g., 60) indicate greater patient confidence in management of medications and therapy relative to a general chronic illness population and lower scores (e.g., 40) indicate lower patient confidence in management of medications and therapy relative to a general chronic illness population. T-scores will be summarized by arm.
Change in Stigma | 6 months
  Change from baseline in stigma will be assessed using the Patient Reported Outcome Measurement Information System Neurological Quality of Life (PROMIS Neuro-QOL) short form questionnaire. The PROMIS Neuro-QOL is an 8-item survey that measures patient-reported perceived disease-related stigma. Responses to each item are scored on a 5-point Likert-like scale ranging from 1 ("Never") to 5 ("Always"). Raw itemized scores are aggregated and transformed to a T-score using a linear transformation. The T-score is centered at 50 with a standard deviation of 10 such that 50 is considered average. Higher scores (e.g., 60) indicate greater perceived stigma relative to a general chronic illness population and lower scores (e.g., 40) indicate lower perceived stigma relative to a general chronic illness population. T-scores will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Rubinstein, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Following publication of main study findings, all collected human subject data will be shared via the NIMH Data Archive (NDA). All collected research data will be uploaded into the Research Domain Criteria Database (RDoC-db) as part of the NDA. The NIMH's guidelines and procedures for sharing data in the RDoC-db specify that raw data be shared on a semiannual basis. To facilitate this process, the study team will use the Research Electronic Data Capture Consortium (REDCap) database to develop an online data management tool where study data can be directly uploaded to the RDoC database.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following the initial upload of raw data as described above, data will be shared in accordance with the standard six-month period for data uploads. All raw data provided will include an NDA Global Unique Identifier and will not include any personally identifiable information. Any analyzed research data expected to be published will be submitted to the NDA no later than the time of publication. Unpublished data will be shared within a year after project completion.
Access Criteria: For access to record-level IPD a Data Access Request must be submitted. Users with NDA credentials may submit Data Access Requests for 1 Permission Group at a time (Broad Use, Controlled Access, or Open Access) from the NDA Permissions Dashboard. Each request includes an NDA Data Use Certification signed by the lead recipient and an authorized Signing Official from recipient's research institution. Additional research staff from the same institution may be added by completing the Senior/Key Person Profile section. All recipients on a Data Use Certification must be affiliated with the recipient's research institution.
  NDA users submitting Data Access Requests for Broad Use and Controlled Access Permission Groups must be sponsored by an NIH recognized institution with a Federalwide Assurance (FWA) and have a research-related need to access NDA data. NDA users submitting Data Access Requests for Controlled Access Permission Groups must adhere to consent-based data use limitations.
URL: https://nda.nih.gov/